CLINICAL TRIAL: NCT02190201
Title: A Randomised Controlled Trial Comparing McGrath Series 5 Videolaryngoscope and Macintosh Laryngoscope for Double Lumen Tube Intubation
Brief Title: Comparison of McGrath and Macintosh Laryngoscope for DLT Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wenlong Yao, M.D., Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJMZK201405001
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Intubation; Difficult; Thoracic Diseases; Intubation Complication
Keywords: videolaryngoscope; double lumen intubation
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- videolaryngoscope (Experimental): DLT intubation with McGrath videolaryngoscope
  Interventions: Device: videolaryngoscope
- Direct laryngoscope (Active Comparator): DLT intubation with Macintosh laryngoscope
  Interventions: Device: Direct laryngoscope

INTERVENTIONS:
Device: videolaryngoscope — a kind of videolaryngoscopes, which are widely used in difficult airways.
  Other Names: McGrath series 5 videolaryngoscope
  Arms: videolaryngoscope
Device: Direct laryngoscope — A kind of traditional laryngoscopes
  Other Names: Macintosh laryngoscopes
  Arms: Direct laryngoscope

SUMMARY:
The investigators previous study showed that McGrath Series 5 videolaryngoscope is an alternative tool for double-lumen tube intubation. But it is not determined about the advantages and disadvantages of McGrath Series 5 videolaryngoscope for double-lumen tube intubation, compared with traditional Macintosh laryngoscope.

DETAILED DESCRIPTION:
The investigators designed a randomised controlled study to compare of McGrath Series 5 videolaryngoscope and Macintosh laryngoscope for DLT intubation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Thoracic surgery required one lung ventilation

Exclusion Criteria:

* Difficult ventilation
* Emergent operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Intubation time | at intubation
  measured with a stopwatch, defined as time from inserting blade to mouth to withdrawal of blade

SECONDARY OUTCOMES:
number of successful intubation at first attempt | at intubation

OTHER OUTCOMES:
Airway evaluation with Cormack-Lehane Score | At intubation
  based on Cormack-Lehane classification. degree 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, M.D., Study Chair — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China